CLINICAL TRIAL: NCT03415906
Title: Influences of Angiotensin-neprilysin Inhibition With Sacubitril/Valsartan (ENTRESTO®) on Centrally Generated Sympathetic Activity in Heart Failure Patients
Brief Title: Influences of Angiotensin-neprilysin Inhibition on Sympathetic Activity in Heart Failure
Acronym: ARNI-Sy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties in recruiting patients
Sponsor: Hannover Medical School (Other)
Collaborators: DLR German Aerospace Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: M17-05-LCZ-ARNI
Record Dates: First submitted 2018-01-02; First posted 2018-01-30 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure
Keywords: angiotensin receptor blocker; neprilysin inhibition; sympathetic activity; baroreflex; microneurography; functional MRI
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan; Angiotensin Receptor Antagonists

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, active-controlled, double-blind, cross-over with randomized sequence of treatments
Who Masked: Participant, Investigator
Masking Description: double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sacubitril+valsartan (Experimental): Combined angiotensin receptor and neprilysin inhibition
  Interventions: Combination Product: sacubitril+valsartan
- valsartan (Active Comparator): Angiotensin receptor inhibition alone
  Interventions: Drug: valsartan

INTERVENTIONS:
Combination Product: sacubitril+valsartan — Combined angiotensin receptor + neprilysin inhibition
  Arms: sacubitril+valsartan
Drug: valsartan — Angiotensin receptor inhibition alone
  Other Names: Angiotensin receptor blocker (AT1-receptor blocker)
  Arms: valsartan

SUMMARY:
The autonomic nervous system plays an important role in controlling the circulation. Increased sympathetic activity has detrimental effects in patients with heart failure.

The purpose of this study is to test the hypothesis that combined angiotensin receptor + neprilysin inhibition results in lower sympathetic activity than angiotensin receptor inhibition alone.

DETAILED DESCRIPTION:
Thirty-five heart-failure patients will be included in a prospective, monocentric, active-controlled, double-blind, cross-over study with randomized sequence of treatments sacubitril+valsartan or valsartan alone. After open-label dose finding and washout patients will be randomly assigned to the treatment sequence [sac+val --> val] or [val --> sac+val]. The two treatment periods of 4 weeks duration will be separated by 2 weeks of washout. At the end of both treatments the state of the cardiovascular system and its control will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Women or men at the age ≥ 18 years, ≤ 80 years and able to give written informed consent
2. Heart failure NYHA class II-III
3. Ejection fraction of 40 % or less
4. Stable dose of an ACE inhibitor or ARB over the last 4 weeks (A 2-day ACE inhibitor washout is scheduled before run-in; see Figure 3 on page 29.)
5. Stable dose of a beta-blocker over the last 4 weeks unless contraindicated or not tolerated
6. Patient has to be in sinus rhythm
7. Patients capable of understanding the investigational nature, potential risks and benefits of the clinical trial
8. Women without childbearing potential defined by:

   * at least 6 weeks after surgical sterilization by bilateral tubal ligation or bilateral oophorectomy or
   * hysterectomy or uterine agenesis or
   * ≥ 50 years and in postmenopausal state ≥ 1 year or
   * < 50 years and in postmenopausal state ≥ 1 year with urine FSH > 40 IU/l and urine estrogen < 30 ng/l or a negative estrogen test OR

   Women of childbearing potential with a negative urine ß-HCG pregnancy test at screening who agree to meet one of the following criteria from the time of screening, during the study and for a period of 7 days following the last administration of study medication:
   * correct use of at least an acceptable effective contraceptive measure. The following are deemed acceptable in this study: hormonal contraceptives (combined oral contraceptives and estrogen-free pills with desogestrel, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release), intrauterine device (IUS))
   * true abstinence (periodic abstinence and withdrawal are not acceptable methods of contraception)
   * sexual relationship only with female partners and/or sterile male partners OR Male
9. Signed written informed consent and willingness to comply with treatment and follow- up procedures.

Exclusion Criteria:

1. History of hypersensitivity or allergy to any of the study drugs, drugs of similar chemical classes, ACE inhibitors (ACE-Is), ARBs, or neprilysin inhibitors, as well as known or suspected contraindications to the study drugs
2. History of angioedema
3. Recent acute decompensated heart failure within 2 months before screening
4. Symptomatic hypotension and/or office systolic BP <110 mmHg at screening measured according to the recommendations of the European Society of Hypertension
5. Combined intake of an ACE inhibitor and ARB over the last 4 weeks
6. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m²
7. Concomitant medication with Aliskiren in patients with Diabetes or patients with eGFR < 60 mL/min/1.73 m²
8. Serum potassium >5.2 mmol/L at Visit 1 (screening)
9. Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid, or other major cardiovascular surgery, PCI, or carotid angioplasty within the 3 months before screening
10. History of heart transplant or on a transplant list or with LV assistance device
11. History of severe pulmonary disease
12. Documented untreated ventricular arrhythmia with syncopal episodes within the 3 months prior to Visit 1
13. Presence of hemodynamically significant mitral and/or aortic valve disease/ left ventricular outflow tract obstruction, except mitral regurgitation secondary to LV dilatation
14. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs
15. Evidence of hepatic disease as determined by any one of the following: aspartate aminotransferase or alanine aminotransferase values exceeding 2× upper limit of normal at Visit 1, history of hepatic encephalopathy, history of esophageal varices, or history of porto-caval shunt
16. Contraindications precluding microneurography measurements, such as relevant peripheral neuropathy as judged by the investigator
17. Pregnancy or lactation period
18. Current participation in any other clinical trial or participation in another clinical trial within 30 days before screening
19. Known or suspected hypersensitivity to any of the active substances or any excipients of the investigational medicinal products
20. Vulnerable subjects (i.e. persons under any administrative or legal supervision or persons kept in detention)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
MSNA burst frequency [bursts/min] | For 5 minutes at the end of both treatments
  Bursts of vasoconstrictor sympathetic nerve activity directed to skeletal muscle (muscle sympathetic nerve activity, MSNA) per minute

SECONDARY OUTCOMES:
DBP [mmHg] | For 5 minutes at the end of both treatments
  Diastolic blood pressure
PVN activity [unitless] | For 20 minutes at the end of both treatments
  Using functional Magnetic Resonance Imaging (fMRI) with concurrent Lower Body Negative Pressure (LBNP), we will identify the paraventricular hypothalamic nucleus (PVN) by its activity change from low to high LBNP stimulation in a 20-minute paradigm. Activity will be reported as a z-scores (no unit) averaged over the entire activation cluster.
NTS activity [unitless] | For 20 minutes at the end of both treatments
  Using functional Magnetic Resonance Imaging (fMRI) with concurrent Lower Body Negative Pressure (LBNP), we will identify the nucleus of the solitary tract (NTS) by its activity change from low to high LBNP stimulation in a 20-minute paradigm. Activity will be reported as a z-scores (no unit) averaged over the entire activation cluster.
MSNA burst incidence [bursts/100 heartbeats] | For 5 minutes at the end of both treatments
  Bursts of vasoconstrictor sympathetic nerve activity normalized to heart rate
MSNA burst area [au/min] | For 5 minutes at the end of both treatments
  Area under the bursts in the integrated neurogram of vasoconstrictor sympathetic nerve activity
Cardiac baroreflex gain [ms/mmHg] | For 5 minutes at the end of both treatments
  Ratio between the changes in ECG RR interval and systolic blood pressure
Sympathetic baroreflex gain [bursts/mmHg] | For 5 minutes at the end of both treatments
  Ratio between the changes in burst frequency and diastolic blood pressure
Sympathetic excitability [bursts] | For 3 minutes at the end of both treatments
  Increase in burst frequency elicited by isometric exercise (handgrip)
NE [nM] | After 20 minutes of supine rest at the end of both treatments
  Venous plasma norepinephrine level

OTHER OUTCOMES:
GLS [%] | For 10 seconds at the end of both treatments
  Echocardiography:
  Global longitudinal strain as assessed using the speckle tracking technique
E/E' [ratio] | For 10 seconds at the end of both treatments
  Echocardiography:
  E = mitral peak velocity of early filling E' = early diastolic mitral annular velocity (mean of E' lateral and E' septal) E and E' are obtained from 3 or 5 heart cycles with sinus rhythm or atrial fibrillation, respectively.
sPAP [mmHg] | For 10 seconds at the end of both treatments
  Echocardiography:
  Systolic pulmonary arterial pressure obtained from 3 or 5 heart cycles with sinus rhythm or atrial fibrillation, respectively.
HR variability [ms²] | For 5 minutes at the end of both treatments
  ECG RR-interval oscillations
BP variability [mmHg²] | For 5 minutes at the end of both treatments
  Blood pressure oscillations
Echocardiographic parameters | For 20 minutes at the end of both treatments
  Cardiac dimension and function as assessed by echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center Hannover, Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Undecided